CLINICAL TRIAL: NCT01625676
Title: Constraint-Induced Aphasia Therapy Following Sub-acute Stroke: A Modified Therapy Schedule
Brief Title: Study of Modified Constraint-Induced Aphasia Therapy Schedule to Treat Patients Following Sub-acute Stroke
Acronym: MCIAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NRZ Magdeburg Median Kliniken GmbH & Co (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIC-2012
Record Dates: First submitted 2012-06-15; First posted 2012-06-21 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Aphasia
Keywords: Aphasia; Rehabilitation of Speech and Language Disorders
MeSH Terms: conditions — Aphasia; Language Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CIAT-Group (Experimental): Patients received a modified constraint-induced therapy schedule
  Interventions: Other: Investigate efficacy of modified ciat schedule
- standard treatment group (Active Comparator): patients received a standard aphasia therapy
  Interventions: Other: examine the efficacy of standard treatment versus modified ciat schedule

INTERVENTIONS:
Other: Investigate efficacy of modified ciat schedule — 2 hours of training over 15 days
  Arms: CIAT-Group
Other: examine the efficacy of standard treatment versus modified ciat schedule — 2 hours of training over 15 days
  Arms: standard treatment group

SUMMARY:
The purpose of this study is to assess the feasibility of modified Constraint-Induced Aphasia Therapy (CIAT) in the early sub-acute stage and to examine the efficacy of modified CIAT versus standard treatment with the same intensity of intervention.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of first-ever stroke
* aphasia in sub-acute stage
* german speakers

Exclusion Criteria:

* presence of residual aphasia
* dysarthria and apraxia of speech

Ages: 34 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-08; Primary Completion 2010-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change of aphasia and aphasic syndromes by Aachen Aphasia Test (AAT) | pretreatment and 4 weeks
change from pretreatment in Aachen Aphasia Test at 8 weeks | pretreatment and 8 weeks
change from pretreatment in Aachen Aphasia Test at 1 year | pretreatment and 1 year

SECONDARY OUTCOMES:
Change of Communicative Activity (CAL) | pretreatment and 4 weeks
change from pretreatment in communication activity (CAL)at 8 weeks | pretreatment and 8 weeks
Change from pretreatment in communication activity (CAL)at 1 year | pretreatment and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Almut A Sickert, PhD, Study Chair — NRZ Median Klinik Magdeburg
Locations (1):
- NRZ Median Klinik, Magdeburg, Germany, Germany

REFERENCES:
- [Derived] Sickert A, Anders LC, Munte TF, Sailer M. Constraint-induced aphasia therapy following sub-acute stroke: a single-blind, randomised clinical trial of a modified therapy schedule. J Neurol Neurosurg Psychiatry. 2014 Jan;85(1):51-5. doi: 10.1136/jnnp-2012-304297. Epub 2013 Jul 4. PMID 23828834